CLINICAL TRIAL: NCT03314103
Title: A Multi-center, Randomized, Double-blinded, Phase 3 Trial to Evaluate the Efficacy Against Herpes Zoster of a Live Attenuated Varicella-Zoster Virus Vaccine in Adults Over 40 Years of Age
Brief Title: Efficacy Trial of a Vaccine to Prevent Herpes Zoster in Adults Over 40 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Principal Investigator, Fengcai Zhu, Profesor, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CS-HZ-2017
Record Dates: First submitted 2017-10-14; First posted 2017-10-19 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): live attenuated varicella-zoster virus vaccine (with live virus >=4.3 LgPFU per dose)
  Interventions: Biological: One shot of the varicella-zoster virus vaccine
- Placebo (Placebo Comparator): Placebo with no live virus
  Interventions: Biological: one shot of placebo

INTERVENTIONS:
Biological: One shot of the varicella-zoster virus vaccine — One shot of the live attenuated varicella-zoster virus vaccine (with live virus >=4.3 LgPFU per dose)
  Arms: Vaccine
Biological: one shot of placebo — one shot of placebo with no live virus
  Arms: Placebo

SUMMARY:
Varicella-zoster virus (VZV) is a herpesvirus that causes two distinct clinical syndromes.Primary infection is manifested as varicella (chickenpox), whereas reactivation of latent VZV results in a localized eruption known as herpes zoster. More than 99.6% of people 40 years of age orolder had evidence of previous VZV infection. This study plans to have 30000 adults 40 years of age or older involoved in a randomized, double-blind, placebo-controlled trial of an investigational live attenuated varicella-zoster virus vaccine. The investigational vaccines are produced by Changchun Changsheng biotechnology co. LTD. The incidence of herpes zoster and the severity, and duration of the associated pain and discomfort were measured after the vaccination. And the safety of the varicella-zoster virus vaccine is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged over 40 years (male or female).
* Able to comply with all clinical trial protocol requirements and willing to complete all the visit plan process during the whole clinical trial observation period.
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able to complete the diary card independently.
* For females only (40-49 years), a negative urine pregnancy test and willing to practice continuous effective contraception during the study.
* Axillary temperature ≤37.0°C.

Exclusion Criteria:

* Prior history of herpes zoster.
* Prior history of vaccination with herpes zoster vaccine or chickenpox vaccine.
* History of allergic disease likely to be exacerbated by any component of the vaccine.
* Taking immunoglobulins and/or any blood products within the last 3 months or will receive these products during the study period.
* Taking certain pharmaceuticals to be like salicylate kind, including aspirin, and difluorosalicylic, or going to take these medicine during the study period.
* Participation in another research study involving receipt of an investigational product in the last 30 days.
* Prior administration of attenuated vaccine in last 28 days.
* Prior administration of subunit vaccine, inactivated vaccine or allergic therapy in last 14 days.
* History of serious disease and the participation in the clinical trial is likely to increase the disease risk and interfere with the observation of clinical trial index.
* Taking immunosuppressive therapy in last 6 months.
* Any autoimmune disease or immunodeficient state, autoimmune disease or immunodeficient disease.
* Active tuberculosis patient.
* Acute or chronic infections at the vaccination day (axillary temperature>37.0°C).
* Coagulation disorders (coagulation factor deficiency, coagulopathy or platelet disorder) diagnosed by doctors, or obvious bruises or blood coagulation noticed.
* Woman who is breast-feeding.
* Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30000 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
The incidence of herpes zoster 30 days after vaccination. | 30 days-2 years after the vaccination
  The incidence of herpes zoster diagnosed in participants 30 days after vaccination.

SECONDARY OUTCOMES:
The incidence of herpes zoster after vaccination. | within 0 day -2 years after the vaccination
  The incidence of herpes zoster diagnosed in participants after vaccination.
The incidence of laboratory-confirmed herpes zoster 30 days after vaccination. | 30 days-2 years after the vaccination
  The incidence of laboratory-confirmed herpes zoster diagnosed in participants 30 days after vaccination.
The incidence of herpes zoster with severe postherpetic neuralgia (ZBPI scores≥3) 30 days after vaccination. | 30 days-2 years after the vaccination
  The incidence of herpes zoster with severe postherpetic neuralgia (ZBPI scores≥3) in participants 30 days after vaccination.
The incidence of herpes zoster with postherpetic neuralgia 30 days after vaccination. | 30 days-2 years after the vaccination
  The incidence of herpes zoster with postherpetic neuralgia in participants 30 days after vaccination.
The incidence of herpes zoster with severe pain (ZBPI scores≥3) 30 days after vaccination. Time Frame: 30 days-2 years after the vaccination | The incidence of herpes zoster with severe pain (ZBPI scores≥3) in participants 30 days after vaccination.
  30 days-2 years after the vaccination
Geometric mean titre, geometric mean fold increase and four-fold increase rate of serum for antibody responses 30 days post-vaccination. | 30 days after the vaccination
  Geometric mean titre, geometric mean fold increase and four-fold increase rate of Serum for antibody responses at day 30 post-vaccination
Geometric mean titre, geometric mean fold increase of serum for antibody responses 6 months post-vaccination. | 6 months after the vaccination
  geometric mean titre, geometric mean fold increase of Serum for antibody responses at 6 months post-vaccination
Geometric mean titre, geometric mean fold increase of serum for antibody responses 12 months post-vaccination. | 12 months after the vaccination
  geometric mean titre, geometric mean fold increase of Serum for antibody responses at 12 months post-vaccination
Geometric mean titre, geometric mean fold increase of serum for antibody responses 24 months post-vaccination. | 24 months after the vaccination
  geometric mean titre, geometric mean fold increase of Serum for antibody responses at 24 months post-vaccination
Occurrence of solicited adverse reactions after the vaccination. | within 14 days after the vaccination
  Occurrence of solicited adverse reactions within 14 days after the vaccination.
Occurrence of adverse reactions after the vaccination. | within 30 days after the vaccination
  Occurrence of adverse reactions within 30 days after the vaccination.
Occurrence of severe adverse reactions after the vaccination. | within 2 years
  Occurrence of severe adverse reactions within 2 years after the vaccination.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hunan Provincial Center for Disease Control and Prevention, Loudi, Hunan
  - Jiangsu Province Centers for Disease Control and Prevention, Nanjing, Jiangsu
  - Zhejiang Provincial Center for Disease Control and Prevention, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No